CLINICAL TRIAL: NCT01186302
Title: Comparison of the Safety, Efficacy, and Feasibility of Medical Abortion Provided by Physicians and Non-physicians in Nepal: a Randomized Controlled, Equivalence Trial.
Brief Title: Comparison of the Safety and Efficacy of Medical Abortion Provided by Physicians and Midlevel Providers in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Health Organization (Other)
Collaborators: Center for Research on Environment, Health and Population Activities (Other)
Responsible Party: Ina Warriner, World Health Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WHO A65550
Record Dates: First submitted 2010-08-20; First posted 2010-08-23 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Medical Abortion
Keywords: medical abortion; Nepal; midlevel providers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midlevel provider (Other): Patients were assigned to a midlevel provider (arm 1) or to a physician (arm 2) for their abortion.
  Interventions: Other: Type of provider
- Physician arm (Other): Patients were assigned to a midlevel provider (arm 1) or to a physician (arm 2) for their abortion.
  Interventions: Other: Type of provider

INTERVENTIONS:
Other: Type of provider — Different types of clinicians have different types of medical training. This study tested whether midlevel providers were as safe and effective in administering medical abortion as doctors. All types of providers underwent the same training in medical abortion and used the same medical abortion regimen.

SUMMARY:
The purpose of the study is to compare the safety, effectiveness, and acceptability of medical abortion provided by doctors and midlevel providers in a developing country where doctors are scarce, such as Nepal. This study is the first to evaluate the independent provision of medical abortion by trained nurses and auxiliary nurse midwives compared to doctors by assessing differences in safety, clinical outcomes, case management decision-making, and acceptability. This study provides scientifically valid data on the administration of medical abortion by midlevel providers working independently in a low-resource, developing country setting. The evidence generated by the study will assist policy makers in developing countries interested in expanding safe abortion services by eliminating the legal requirement limiting prescription of medical abortion to doctors where medical abortion is not restricted by law.

DETAILED DESCRIPTION:
Each year, some 210 million women throughout the world become pregnant and nearly one in five chooses to terminate the pregnancy (Singh et al., 2009). Approximately, 22 million pregnancies are terminated unsafely; of these, the vast majority (98%) take place in developing countries (WHO, Forthcoming). Access to safe abortion services is a challenge for many women with unwanted pregnancies in developing countries because of restrictive legislation, a shortage of skilled staff or other barriers.

Non-surgical methods of abortion, known as medical abortion, have been developed that use safe and effective drug-based methods for induced abortion. Prescribing authority is generally limited to doctors, however. As a result, medical abortion remains under-utilized and is often inaccessible for many women in developing countries seeking public sector providers trained in medical abortion in areas where there are no doctors.

Midlevel providers (non-physician clinicians such as nurses and midwives) have the potential to provide accessible, low-cost, and safe abortion services in many countries, especially in the developing world. They are more cost-effective to employ than doctors and often work in areas where doctors are in short supply, providing much needed health services to under-served areas while conserving resources. Training midlevel providers in the independent provision of medical abortion with appropriate referral systems would expand access to safe abortion services to lower levels of the health care system where there is no doctor and complement a global health systems trend towards task-shifting where doctors are costly and scarce (WHO, 2007).

The overall objective of the study is to obtain evidence on the safety and effectiveness of medical abortions performed by government trained and certified midlevel providers and physicians to inform policy makers interested in or committed to expanding and decentralizing medical abortion services.

ELIGIBILITY:
Inclusion Criteria:

* Before randomization: Gestational age not more than 63 days as estimated by last menstrual period (LMP).
* After randomization: Gestational age not more than 63 days as estimated by abdominal and bimanual pelvic examination.
* Above national age of consent
* Willing to return to the clinic for misoprostol on Day 3 and for a follow-up visit on Day 10 to 14.
* Residence within the geographical area specified for each clinic and no more than one hour from emergency referral services.
* Willing to provide written informed consent to participate in the study and to be randomly assigned to a provider team.
* Able to understand the nature of the study, advice and instructions given by health providers.

Exclusion Criteria:

* Previous allergic reaction to one of the drugs in the medical abortion regimen
* Known or suspected ectopic pregnancy or undiagnosed adnexal mass
* Inherited porphyria (rare genetic blood diseases)
* Chronic adrenal failure
* Long term corticosteroid therapy
* Haemorrhagic disorder or anticoagulant therapy (blood thinner medications)
* IUD in utero that can not be removed before taking mifepristone
* Previous enrolment in the study (i.e. no repeat abortions; only one abortion per woman in the study)
* Unwilling or unable to return to clinic for follow-up visit.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1104 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Complete abortion | 30 days
  The primary outcome measure was a successful (complete) abortion, defined as no ongoing pregnancy at clinical examination and no surgical intervention necessary.

SECONDARY OUTCOMES:
Complications from medical abortion | 30 days
  Defined as life-threatening events requiring hospitalization: haemorrhage requiring a blood transfusion, hospitalization (iv fluids, iv antibiotics), or laparatomy for ectopic pregnancies.

CONTACTS AND LOCATIONS:
Overall Officials: Kusum Thapa, MD, Principal Investigator — Department of Obstetrics and Gynaecology, Paropakar Maternity and Women Hospital (Maternity Hospital), Kathmandu, Nepal; Ina Warriner, PhD, Study Director — World Health Organization
Locations (1):
- Center for Research and Environmental Health and Population Activities (CREHPA), Kathmandu, Nepal

REFERENCES:
- [Background] Warriner IK, Meirik O, Hoffman M, Morroni C, Harries J, My Huong NT, Vy ND, Seuc AH. Rates of complication in first-trimester manual vacuum aspiration abortion done by doctors and mid-level providers in South Africa and Vietnam: a randomised controlled equivalence trial. Lancet. 2006 Dec 2;368(9551):1965-72. doi: 10.1016/S0140-6736(06)69742-0. PMID 17141703
- [Derived] Tamang A, Shah IH, Shrestha P, Warriner IK, Wang D, Thapa K, My Huong NT, Meirik O. Comparative satisfaction of receiving medical abortion service from nurses and auxiliary nurse-midwives or doctors in Nepal: results of a randomized trial. Reprod Health. 2017 Dec 16;14(1):176. doi: 10.1186/s12978-017-0438-7. PMID 29246235
- [Derived] Warriner IK, Wang D, Huong NT, Thapa K, Tamang A, Shah I, Baird DT, Meirik O. Can midlevel health-care providers administer early medical abortion as safely and effectively as doctors? A randomised controlled equivalence trial in Nepal. Lancet. 2011 Apr 2;377(9772):1155-61. doi: 10.1016/S0140-6736(10)62229-5. PMID 21458058